CLINICAL TRIAL: NCT01941433
Title: Proof of Concept Study of the Arthritis Health Journal, a Patient Passport for Rheumatoid Arthritis
Brief Title: Arthritis Health Journal Proof of Concept Study
Acronym: AHJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Initiative for Outcomes in Rheumatology Care (Other); Vancouver Coastal Health (Other Government); Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Diane Lacaille, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H12-00691
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; self-management; online; patient passport
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthritis Health Journal (Experimental): Participants in this group will use the Arthritis Health Journal in the first 6 months of study.
  Interventions: Behavioral: Arthritis Health Journal
- Control (Other): Participants in this group will receive a delayed intervention. They will receive usual care for the first 6 months of study, during which time they will contribute control data, and they will use the Arthritis Health Journal in the second 6 months of study, during which time they will contribute intervention data.
  Interventions: Behavioral: Arthritis Health Journal

INTERVENTIONS:
Behavioral: Arthritis Health Journal

SUMMARY:
The purpose of this study is to determine whether an online patient passport tool called the Arthritis Health Journal can assist people with rheumatoid arthritis in managing their disease.

DETAILED DESCRIPTION:
Patient passports have been developed and used in chronic diseases, such as diabetes, to promote active involvement of patients in their care, and have led to better treatment and health outcomes. In rheumatoid arthritis (RA), active involvement of patients in monitoring their symptoms and their disease activity may facilitate treatment according to current recommendations, which emphasize the need for aggressive treatment to suppress inflammation and for using a "Treat to Target" approach where treatment is escalated until a target is reached and is promptly modified when target is no longer met. In this study, the investigators have developed an online tool that aims to help people with RA monitor their symptoms and their disease activity and self-manage their arthritis. The investigators will perform a proof of concept study assessing how the Arthritis Health Journal affects consumer effectiveness, patient self-efficacy, communication with health professionals, shared decision-making, and satisfaction with medical care. The investigators will also evaluate the feasibility and satisfaction with using the Arthritis Health Journal. The investigators will use a stepped wedge study design, in which 50 participants will be randomized to either the intervention group (immediate use of the Arthritis Health Journal) or the control group (waitlisted for 6 months). Due to the nature of the intervention, the study is not blinded.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Have a diagnosis of rheumatoid arthritis
* Be under the ongoing care of a rheumatologist
* Be comfortable using a computer and online applications
* Have access to an Internet connection
* Be able to read and write English without needing a translator

Exclusion Criteria:

* Younger than 18 years of age;
* Diagnoses of arthritis other than rheumatoid arthritis
* not under the ongoing care of a rheumatologist
* not comfortable using a computer
* lack of Internet access
* inability to read and write in English without a translator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Self-Management Behaviours | 6 months
  We will use the overall score from the Partners in Health Scale, an 11 item questionnaire based on the principles of self-management, which measures people's ability to engage in behaviours for the self-management of a chronic disease.

SECONDARY OUTCOMES:
Self-Efficacy | 6 months
  We will use the Stanford Self-Efficacy Scale to measure patient's confidence in their ability to perform certain actions to manage their disease and cope with the consequences of their disease. Specifically we will include the "Manage Arthritis Symptoms", "Manage Disease in General", and "Communicate with Physician" subscales.
Consumer Effectiveness | 6 months
  We will use the Effective Consumer (EC-17) scale to measure patient's ability to deal with a chronic condition and make decisions about their health care. We will use the global EC-17 score, as well as results to individual questions (6, 7, 9, and 13) which were selected for their relevance to our intervention.
Patient Satisfaction with Care | 6 months
  We will use the Patient Satisfaction Questionnaire to measure satisfaction with care and patient-physician interactions.
Self-Management Behaviours | 6 months
  We will measure the results of individual questions 7 to 11 from the Partners in Health Scale, which specifically measure involvement in aspects of care relevant to our intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Lacaille, MD MHSc, Principal Investigator — Arthritis Research Centre of Canada
Locations (1):
- Arthritis Research Centre of Canada, Richmond, British Columbia, Canada